CLINICAL TRIAL: NCT06853275
Title: The Influence of Movement Velocity Biofeedback on Muscle Activation and Self Perception in Older Adults With Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Foundation for Physical Therapy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2005068
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sarcopenia; Sarcopenia in Elderly; Age-associated Muscle Loss
Keywords: Geriatrics; Neuromuscular; Rehabilitation; Sarcopenia; Velocity-based training
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Focus (Experimental)
  Interventions: Behavioral: Experimental: External Focus
- Internal Focus (Other)
  Interventions: Behavioral: Other: Internal Focus

INTERVENTIONS:
Behavioral: Experimental: External Focus — Participants will perform a short, standardized warm-up (1 set of 10 repetitions of 20% of the participant's estimated 1-repetition maximum). Following the warm-up, participants will perform 30 repetitions using 50% of their estimated 1-repetition maximum on a leg press machine. Participants will receive visual feedback from a linear position transducer for each repetition, indicating the speed of the last repetition/movement.
  Arms: External Focus
Behavioral: Other: Internal Focus — Arm Description: Participants will perform a short, standardized warm-up (1 set of 10 repetitions of 20% of the participant's estimated 1RM). Following the warm-up, participants will perform 30 repetitions using 50% of their estimated 1-repetition maximum on a leg press machine. Participants will NOT receive visual feedback for each repetition. This is the control condition.
  Arms: Internal Focus

SUMMARY:
The overall objective for this clinical trial is to provide evidence for internal and external cueing for physical therapists and other rehabilitation clinicians to optimize resistance training within rehabilitation for older adults. The main questions it aims to answer are:

* What is the impact of external focus (providing velocity of movement for each repetition) compared to internal focus (i.e., no cues, control group) on physical percent velocity loss and neuromuscular activation in older adults with sarcopenia?
* Does internal and external focus influence motivation and perceptual workload following resistance training in older adults with sarcopenia?

Researchers will compare external focus to internal focus to see if external focus impacts percent velocity loss, motivation, and perceived workload.

Participants will:

* Visit the lab once per week for 3 weeks
* Perform exercise testing using a leg press
* Answer questionnaires regarding perceived workload and motivation before and after exercise

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults 60-95 years of age
* Physically independent
* Free of severe mental impairment
* Score 4 or greater on the SARC-F sarcopenia questionnaire

Exclusion Criteria:

* Participated in a structured resistance training program in the last 12 months
* Had a lower extremity injury or surgical intervention within the past 6 months
* Have neuromuscular (i.e., Parkinson's Disease, Multiple Sclerosis), circulatory, or edema pathology

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Velocity Loss | Week 1 and Week 2 Timepoints
  The linear position transducer is a spring-powered retractable apparatus that attaches to the leg press on one end and to the machine near the participant's hip joint. Velocity data from a linear position transducer will be collected following each repetition. Percent velocity loss (%VL) measures the reduction in the movement speed from the initial repetition to the final repetition. The %VL will quantify the level of fatigue and performance decline that occurs throughout the repetitions of leg press. This would suggest that a higher %VL would indicate a greater degree of fatigue, while a lower %VL loss would indicate a better ability to maintain movement velocity across the repetitions.
Muscle Activation | Baseline, Week 1, and Week 2 Timepoints
  To examine muscle activation, surface electromyographic (sEMG) signals will be collected in millivolts (mV) during each repetition using wireless sEMG sensors from the right vastus lateralis. A higher number of millivolts is associated with greater muscular activation. All sEMG signals will use a commercially available signal acquisition system. To optimize signal quality, the skin will be prepared, and the surface electrodes will be secured to the skin with skin-sensor adhesive in a standardized position directly above the muscle in line with the muscle fiber pennation in a bipolar fashion. An electrogoniometer will be placed across the right knee's joint space. The electrogoniometer will be calibrated to 90° flexion and 180° full extension of the knee joint.
Motivation | Week 1 and Week 2 Timepoints
  The Dundee Stress State Questionnaire (DDSQ) has been used to determine task stress and performance impact of stress on task completion. Our proposal focuses on the motivation construct (15 item questionnaire, ~5 minutes to complete) of the DDSQ which has been shown to be reliable and scored on a 4-point Likert scale (Extremely = 4 Very much = 3 Somewhat = 2 A little bit = 1 Not at all = 0). The maximum score possible is 60 points and minimum score possible is 0 points. Higher scores indicate higher motivation. Note that certain items are reverse coded when scoring. Motivation will be assessed before sessions to determine baseline motivation to complete the resistance training protocol and 10 minutes after the resistance training protocol to determine if the visual movement velocity biofeedback improves motivation throughout the resistance training protocol.
Perceived Workload | Week 1 and Week 2 Timepoints
  Perceived workload will be assessed using the NASA task index (NASA-TLX). This questionnaire assesses six separate indices that examine the mental demand, physical demand, temporal demand, performance, effort, and frustration level following the completion of the resistance training protocol. Adjusted scores range from 0-500 with higher scores indicate greater demand, failure, higher effort, or higher frustration. The NASA-TLX will provide valuable information about how visual movement velocity biofeedback may change the perceived workload compared to the non-biofeedback condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data will be housed in the Creighton Digital Repository. Sharing beyond this registry will be handled on a case-by-case basis.